CLINICAL TRIAL: NCT01642823
Title: Cancer Biology of Retinoblastoma
Status: Terminated | Type: Observational
Why Stopped: Logistics
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: PEDSEYE0002
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Retinoblastoma
Keywords: retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — retinoblastoma tumor tissue sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- retinablastoma tumor tissue

SUMMARY:
Many children with the childhood cancer, Retinoblastoma, have surgery to remove the tumor and sometimes the entire eye. The purpose of this study is to collect the extra tissue from patients who undergo tumor removal for laboratory experiments that will help us understand not only what occurs in retinoblastoma cells but also how cells normally function. Some of these studies will include an evaluation of how cells control the way that genes are expressed, how cells "know" to become retinal cells, how cells remain retinal cells, how cells lose their identity as retinal cells, what changes make retinoblastoma cells different from normal retinal cells, and what changes make some retinoblastomas worse than others.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have retinoblastoma
* Patient must be receiving biopsy, partial surgical excision of the tumor, complete excision of the tumor, or enucleation of the eye as part of their standard care.
* Parental consent

Exclusion Criteria:

* Diagnosis other than Retinoblastoma
* No surgical sampling of tumor is planned as part of standard care
* Parental preference to not participate.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Retinoblastoma patients undergoing surgical removal of part or all of their tumor, with or without the remainder of the eye
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Change in efficiency of reprogramming in cells with "naturally occurring" retinoblastoma mutations | After appropriate time, e.g., 7, 10, 14 days after reprogramming
  Comparison of number of reprogramming events (defined by colony formation assay and normalized for number of cell plated) as well as the time to reprogramming.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Sage, Principal Investigator — Stanford University
Locations (2):
- Stanford University Cancer Institute, Stanford, California, United States
- Unidad Nacional de Oncologia Pediatrica, Guatemala City, Guatemala